CLINICAL TRIAL: NCT03716557
Title: A Prospective Single Blind Pilot Study to Investigate the Dynamic Brain Imaging Response to Changes in Frequency Parameters in Patients With Spinal Cord Stimulation With Intractable Neuropathic Pain
Brief Title: A High Frequency Spinal Cord Stimulation PET-CT Scan Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 011768
Record Dates: First submitted 2018-10-22; First posted 2018-10-23 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Neuropathic Pain
Keywords: spinal cord stimulation; high frequency stimulation; paraesthesia-free
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Single-blind crossover design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal Cord Stimulation 4000Hz (Experimental): Patients will trial Spinal Cord Stimulation 4000Hz for 4 weeks. PET/CT scan will be conducted at the end of this period.
  Interventions: Device: Spinal Cord Stimulation 4000Hz
- Spinal Cord Stimulation 10000Hz (Experimental): Patients will trial Spinal Cord Stimulation 10,000Hz for 4 weeks. PET/CT scan will be conducted at the end of this period.
  Interventions: Device: Spinal Cord Stimulation 10000Hz
- Spinal Cord Stimulation 40Hz (Active Comparator): Patients will trial Spinal Cord Stimulation 10,000Hz for 4 weeks. PET/CT scan will be conducted at the end of this period.
  Interventions: Device: Spinal Cord Stimulation 40Hz

INTERVENTIONS:
Device: Spinal Cord Stimulation 4000Hz — Differential programming of the Boston Scientific Precision™ Plus Spinal Cord Stimulator System
  Arms: Spinal Cord Stimulation 4000Hz
Device: Spinal Cord Stimulation 10000Hz — Differential programming of the Boston Scientific Precision™ Plus Spinal Cord Stimulator System
  Arms: Spinal Cord Stimulation 10000Hz
Device: Spinal Cord Stimulation 40Hz — Differential programming of the Boston Scientific Precision™ Plus Spinal Cord Stimulator System
  Arms: Spinal Cord Stimulation 40Hz

SUMMARY:
This study aims to investigate the clinical response to Spinal Cord Stimulation frequency parameters: 40Hz, 4000Hz and 10000Hz and explore the brain imaging changes using PET-CT scans. The response to these stimulator settings on health related quality of life will also be measured using validated questionnaires.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is a treatment option for people suffering with chronic neuropathic back and leg pain. Conventionally, patients receiving SCS are provided with tonic stimulation parameters, where the frequency of electrical pulses is set at 40-60Hz. The major side effect of tonic SCS parameters is the onset of paraesthesia, a tingling or pins and needles sensation within the target region, which can cause discomfort for some patients. However, newer methods include high-frequency stimulation (HF) which is able to provide paraesthesia free stimulation, ultimately providing better patient tolerability. HF stimulation is widely offered to patients with SCS as part of routine clinical practice. However, the effect on pathways in the brain remains to be characterised. This study therefore aims to investigate the clinical response to three frequency parameters 40Hz, 4000Hz and 10000Hz and also explore the brain imaging changes using PET-CT scans. The response to these stimulator settings on health related quality of life will also be measured using validated questionnaires.

20 patients who are deemed suitable for SCS as part of NICE guidelines 159 pathway will be recruited for the study. All patients will have a baseline PET-CT scan and undergo first stage of SCS where they will be offered tonic 40Hz settings as part of trial stimulation. If successful (>50% improvement in pain scores) patients will be offered second stage and continue to receive 40Hz stimulation for 4 weeks. After a second PET-CT scan they are randomised to receive either 4000Hz or 10000Hz stimulation for 4 more weeks, then cross-over treatment for another 4 weeks. PET-CT scans will be performed between each level of stimulation and at the end of the study (4 in total).

ELIGIBILITY:
Inclusion Criteria:

* Patients with intractable lumbar neuropathic pain who are due to receive Percutaneous Spinal Cord Stimulation as part of their standard treatment per NICE HTA guidance 159 at Barts Health NHS Hospitals.
* Patients between 18 and 75 years of age.
* Patients who have given their written informed consent.
* Female patients of childbearing potential must be using adequate contraception (i.e. using oral or IM contraception or an IUCD) and must have a negative urine pregnancy test.
* Patients must be able to communicate in English in order to complete validated questionnaires written in English only.

Exclusion Criteria:

* Patients with diabetes or any underlying neurological condition.
* Patients known to have a condition that in the investigator's judgement precludes participation in the study.
* Patients who have received an investigational drug or have used an investigational device in the 30 days preceding study entry.
* Patients unable to comply with the study assessments and to complete the questionnaires.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
The change in patient reported back pain levels (Numerical Rating Score) | Baseline, 4-weeks post implant, 4-weeks post randomisation, 4-weeks post crossover
  The Numerical Rating Scale will be used to measure patient reported pain levels. The scale is from 0 (no pain) to 10 (extreme pain).

SECONDARY OUTCOMES:
PET/CT Scans | Baseline, 4-weeks post implant, 4-weeks post randomisation, 4-weeks post crossover
  Investigate the changes in the brain following Spinal Cord Simulator (SCS) programmed with the various settings (frequency: 40Hz, 4000Hz and 10000Hz) using imaging technology (PET-CT scan)
Oswestry Disability Index (ODI) | Baseline, 4-weeks post implant, 4-weeks post randomisation, 4-weeks post crossover
  A low back pain functional disability outcome tool. The final score ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound.
Patients Global Impression of Change (PGIC) | Baseline, 4-weeks post implant, 4-weeks post randomisation, 4-weeks post crossover
  A scale to measure the patient's belief about the efficacy of treatment. The scale is from 1 (no change) to 7 (a great deal better). Higher PGIC scores are associated with greater improvement in pain.
EQ-5D-5L | Baseline, 4-weeks post implant, 4-weeks post randomisation, 4-weeks post crossover
  A standardised measure of health status. A summary index with a maximum score of 1 can be derived from five questions. The maximum score of 1 indicates the best health state. There is also a visual analogue scale (0-100) to indicate the general health status with 100 indicating the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, MD, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poply K, Haroon A, Ganeshan B, Nikolic S, Sharma S, Ahmad A, Ellamushi H, Parsai A, Mehta V. Dynamic Brain Imaging Response to Spinal Cord Stimulation Differential Frequencies DiFY SCS-PET Clinical Trial. Neuromodulation. 2023 Jul;26(5):988-998. doi: 10.1016/j.neurom.2022.07.012. Epub 2022 Sep 21. PMID 36151010